CLINICAL TRIAL: NCT00095342
Title: A Double-Blind, Placebo-Controlled, Parallel, Randomized Study to Evaluate the Efficacy and Safety of 3 Oral Dose Levels of TMI-005 in Subjects With Active Rheumatoid Arthritis on a Background of Methotrexate
Brief Title: Study Evaluating TMI-005 in Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3140A1-200
Record Dates: First submitted 2004-11-02; First posted 2004-11-03 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — apratastat

INTERVENTIONS:
Drug: TMI-005

SUMMARY:
The primary objective of this clinical research study is to compare the efficacy and the safety of 3 dose levels of oral TMI-005 in comparison with placebo in subjects with active Rheumatoid Arthritis (RA) who have been receiving stable doses of Methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

* Meet American College of Rheumatology (ACR) criteria for RA
* Have active RA
* Disease duration of at least 6 months
* Disease onset at > 16 years of age.

Exclusion Criteria:

* Any prior use of anti-TNF alpha biologics, rituximab, receipt of anti-CD4 or diphtheria interleukin-2 fusion protein or other immunosuppressive biologics (except for anakinra)
* Largely or wholly incapacitated with the subject bedridden or confined to a wheelchair, permitting limited or no self-care
* Pregnant or breastfeeding women or women planning to become pregnant during the study or within 12 weeks after the last dose of test article

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (8):
- United States (4):
  - Indianapolis, Indiana
  - Syracuse, New York
  - Duncansville, Pennsylvania
  - West Reading, Pennsylvania
- Canada (4):
  - Montreal, Quebec
  - Ste-Foy, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan